CLINICAL TRIAL: NCT03775369
Title: Influence of Physical Activity in Patients With High Grade Glioma (WHO III° and IV°) on Patients' Psychological Well Being, Sleep and Quality of Life
Brief Title: Glioma and Exercising
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University Basel, Department of Sport, Exercise and Health, Division of Sport Science and Psychosocial Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-01314; ch18Cordier
Record Dates: First submitted 2018-12-04; First posted 2018-12-13 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: High Grade Glioma
Keywords: interventions of physical activity and exercising (PAE); resistance training; endurance training
MeSH Terms: conditions — Glioma | interventions — Endurance Training; Counseling; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Endurance training (Active Comparator): Endurance Training (warm-up; endurance on bike; brisk walking; cooling down; group sessions; supervised; moderate and individualized exercising load):
  6 weeks, 2 sessions/week, 40-60min/session
  Interventions: Other: endurance training
- Resistance training (Active Comparator): Resistance Training (warm-up; resistance training units; cooling down; group sessions; supervised; moderate and individualized exercising load):
  6 weeks, 2 sessions/week, 40-60min/session
  Interventions: Other: resistance training
- Control condition (Active Comparator): Control condition (individualized counselling, but not intended as a bona fide intervention, that is to say: not intended to actively improve participants' well-being):
  6 weeks, social support and counseling,1-2 sessions/week; 30 min/session
  Interventions: Other: social support and counseling

INTERVENTIONS:
Other: endurance training — physical activity and exercising (PAE)
  Arms: Endurance training
Other: social support and counseling — social support and counseling
  Arms: Control condition
Other: resistance training — physical activity and exercising (PAE)
  Arms: Resistance training

SUMMARY:
To investigate the influence of two physical activity and exercising (PAE) interventions, namely resistance training and endurance training in relation to quality of life, depression, fatigue, sleep, anxiety, stress and coping, body image, and social interactions (psychological dimensions); cardiorespiratory fitness, morning cortisol secretion, inflammatory markers, and objective sleep (physiological dimensions), along with cancer-related dimensions

DETAILED DESCRIPTION:
Patients with high grade glioma (WHO III° and IV°) and undergoing radiotherapy, chemotherapy, or both radio- and chemotherapy suffer from decreased quality of life (QoL). This study is to analyse the influence of two adjuvant interventions of physical activity and exercising (PAE) (namely resistance training and endurance training) in relation to quality of life, depression, fatigue, sleep, anxiety, stress and coping, body image, and social interactions (psychological dimensions); cardiorespiratory fitness, morning cortisol secretion, inflammatory markers, and objective sleep (physiological dimensions).

ELIGIBILITY:
Inclusion Criteria:

* Patients with high grade glioma (WHO III° and IV°), and undergoing radiotherapy, chemotherapy, or both
* Willing and able to follow the study intervention
* Signed written informed consent

Exclusion Criteria:

* Severe psychiatric (psychosis, suicidal behavior, substance use disorder) and somatic comorbidities (severe cardiovascular disease, severe diabetes, impairments of the musculo-skeletal system)
* patients not willing or able anymore to follow the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Functional Assessment of Cancer Therapy Scale (FACT) | Baseline and week 3 and week 6
  Cancer-related Quality of Life (QOL) assessed by Functional Assessment of Cancer Therapy Scale (FACT), a self-report instrument which measures multidimensional QOL. The FACT evaluation system uses a 29-49 item compilation of a generic core and numerous subscales (9-20 items each) which reflect symptoms associated with different diseases, symptom complexes and treatments.
Change in Hamilton Depression Rating Scale (HDRS) | Baseline and week 3 and week 6
  HDRS scale to assess patients' severity of Depression (mood, feelings of guilt, suicide ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms); each item on the questionnaire is scored on a 3 or 5 point scale; a score of 0-7 is considered to be normal
Change in Intolerance of Uncertainty Scale (IU) | Baseline and week 3 and week 6
  IU: 5-point rating scale (1 = not at all characteristic of me, 5 = entirely characteristic of me) indicating how much patient agrees with the item. The higher the overall score is, the more the respondent is assumed to be more intolerant of uncertainty
Change in Insomnia Severity Index (ISI) | Baseline and week 3 and week 6
  ISI is a 7-item screening measure for insomnia. Items answered on 5-point rating scales (0 = not at all, 4 = very much)
Change in Perceived Stress Scale (PSS) | Baseline and week 3 and week 6
  General perceived stress is assessed with the 10-item Perceived Stress Scale (PSS). The PSS measures the degree to which respondents find their lives unpredictable, uncontrollable and overloading. Answers were given on a five-point Likert-type scale anchored at 1 (never) to 5 (very often). Four items were reverse scored. The mean was calculated in order to obtain an overall score.
Change in Fatigue Severity Scale | Baseline and week 3 and week 6
  nine items, and answers are given on seven-point rating scales ranging from 1 (not at all) to 7 (definitively/almost always), with higher mean scores reflecting greater fatigue
Change in Mental Toughness Questionnaire (MTQ48) | Baseline and week 3 and week 6
  The 48 item MTQ48 measures the subcomponents challenge, commitment, emotional and life control, and interpersonal confidence and confidence in ability. Answers are given on five-point Likert-type scales ranging from 1 (=strongly disagree) to 5 (=strongly agree), with higher scores reflecting greater MT
Change in International Physical Activity Questionnaire | Baseline and week 3 and week 6
  questionnaire consists of several items and asks about the amount of days with walking, moderate and vigorous physical activity.
Change in submaximal 6-min walking test (6MWT) | Baseline and week 3 and week 6
  To assess functional exercise capacity, distance walked during 6 min will be assessed and compared to reference age and gender norms
Change in Grip force | Baseline and week 3 and week 6
  Maximum isometric grip force of the dominant hand is assessed using the hand dynamometer. Participants make three attempts. Mean outcomes is compared to reference data

SECONDARY OUTCOMES:
Change in sleep continuity assessed by EEG | Baseline and week 6
  Sleep is objectively assessed via an easy-to-use in-home sleep-EEG. It consists of three electrodes and measures sleep continuity (awakenings after sleep onset: number of duration of awakenings)
Change in C reactive protein (CRP) (mg/l) | Baseline and week 6
  blood samples are taken before and after the 6MWT and grip force test to assess inflammatory marker CRP (mg/l)
Change in sleep architecture (min; %) | Baseline and week 6
  Sleep is objectively assessed via an easy-to-use in-home sleep-EEG. It consists of three electrodes and measures sleep architecture (wake, Non-rapid eye movement (REM)- sleep stages 1-4 (min; %); REM-sleep (min; %).

CONTACTS AND LOCATIONS:
Overall Officials: Serge Brand, PD Dr. phil, Principal Investigator — Department of Sport, Exercise, and Health, University of Basel
Locations (2):
- Switzerland (2):
  - University Hospital Basel, Department of Neurosurgery, Basel
  - Department of Sport, Exercise and Health, University of Basel, Basel

REFERENCES:
- [Derived] Cordier D, Gerber M, Brand S. Effects of two types of exercise training on psychological well-being, sleep, quality of life and physical fitness in patients with high-grade glioma (WHO III and IV): study protocol for a randomized controlled trial. Cancer Commun (Lond). 2019 Aug 9;39(1):46. doi: 10.1186/s40880-019-0390-8. PMID 31399142